CLINICAL TRIAL: NCT07216482
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Enlicitide Decanoate Coadministered With Rosuvastatin in Adults With Hyperlipidemia
Brief Title: A Clinical Study of Enlicitide in Participants With High Cholesterol (MK-0616-037)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 0616-037; U1111-1319-9502 (Registry Identifier: UTN); 2025-521495-54-00 (Registry Identifier: EU CT); MK-0616-037 (Other: MSD)
Record Dates: First submitted 2025-10-10; First posted 2025-10-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — MK-0616; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Enlicitide (Experimental): Participants will receive enlicitide and a rosuvastatin-matching placebo. Both will be delivered orally once daily (QD) for up to 12 weeks.
  Interventions: Drug: Enlicitide; Drug: Placebo for Rosuvastatin
- Enlicitide + Rosuvastatin (Experimental): Participants will receive enlicitide and rosuvastatin. Both will be delivered orally QD for up to 12 weeks.
  Interventions: Drug: Enlicitide; Drug: Rosuvastatin
- Rosuvastatin (Active Comparator): Participants will receive rosuvastatin and an enlicitide-matching placebo. Both will be delivered orally QD for up to 12 weeks.
  Interventions: Drug: Rosuvastatin; Drug: Placebo for Enlicitide
- Placebo (Placebo Comparator): Participants will receive an enlicitide-matching placebo and a rosuvastatin-matching placebo. Placebos will be delivered orally QD for up to 12 weeks.
  Interventions: Drug: Placebo for Enlicitide; Drug: Placebo for Rosuvastatin

INTERVENTIONS:
Drug: Enlicitide — Oral Tablet
  Other Names: MK-0616; Enlicitide decanoate
  Arms: Enlicitide; Enlicitide + Rosuvastatin
Drug: Rosuvastatin — Oral Capsule
  Arms: Enlicitide + Rosuvastatin; Rosuvastatin
Drug: Placebo for Enlicitide — Oral Tablet
  Arms: Placebo; Rosuvastatin
Drug: Placebo for Rosuvastatin — Oral Capsule
  Arms: Enlicitide; Placebo

SUMMARY:
Researchers designed a study medicine called enlicitide to lower low-density lipoprotein cholesterol (LDL-C). In this study, researchers want to learn about giving enlicitide with another medicine called rosuvastatin. Rosuvastatin is a standard (usual) treatment to lower LDL-C.

The goal of this study is to learn if enlicitide given with rosuvastatin works better than placebo on lowering LDL-C in a person's blood. A placebo looks like the study medicine but has no study medicine in it. Using a placebo helps researchers better understand the effects of a study medicine.

ELIGIBILITY:
Inclusion Criteria:

-Has either not received lipid-lowering therapy (LLT) or has not received certain LLTs within a specified time period prior to the study.

Exclusion Criteria:

* Has a history of homozygous familial hypercholesterolemia (FH), compound heterozygous FH, or double heterozygous FH.
* Had a heart failure hospitalization within 3 months before Screening.
* Is unwilling to take a statin, and/or has a history of statin-associated muscle symptoms or other statin-related AEs to any statin and dose, and/or is known to be intolerant to 1 or more statins.
* Has a history of any of the following conditions: (1) Myopathy, myositis, rhabdomyolysis, or unexplained muscle pain; (2) Muscular or neuromuscular disease; (3) Neuropathy, fibromyalgia, or chronic pain; or (4) Has a personal or family history of hereditary muscular disorders.
* Has active or chronic hepatobiliary or hepatic disease.
* Has known human immunodeficiency virus (HIV) infection.
* Is undergoing or previously underwent an LDL-C apheresis program within 3 months before Screening or plans to initiate an LDL-C apheresis program.
* Has received any medication that may interact with rosuvastatin within 5 half-lives prior to Screening or is planning to initiate such treatment.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 975 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2026-12-02 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Mean Percent Change from Baseline in LDL-C at Week 8 (Enlicitide + Rosuvastatin Versus Placebo) | Baseline and Week 8
  Blood samples will be collected at baseline and at Week 8 to assess mean percent change in LDL-C between participants treated with enlicitide and rosuvastatin versus placebo.

SECONDARY OUTCOMES:
Mean Percent Change from Baseline in LDL-C at Week 8 | Baseline and Week 8
  Blood samples will be collected at baseline and at Week 8 to assess mean percent change in LDL-C.
Mean Percent Change from Baseline in Apolipoprotein B (ApoB) at Week 8 | Baseline and Week 8
  Blood samples will be collected at baseline and at Week 8 to assess mean percent change in ApoB.
Number of Participants with One or More Adverse Events (AEs) | Up to approximately 20 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants who Discontinue Study Drug Due to One or More AEs | Up to approximately 12 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Mean Percent Change from Baseline in LDL-C at Week 12 | Baseline and Week 12
  Blood samples will be collected at baseline and at Week 12 to assess mean percent change in LDL-C.
Mean Percent Change from Baseline in Non-High-Density Lipoprotein Cholesterol (non-HDL-C) at Week 8 | Baseline and Week 8
  Blood samples will be collected at baseline and at Week 8 to assess mean percent change in non-HDL-C.
Percent Change from Baseline in Lipoprotein (a) (Lp[a]) at Week 8 | Baseline and Week 8
  Blood samples will be collected at baseline and at Week 8 to assess percent change in Lp(a).
Percentage of Participants with LDL-C <70 mg/dL and ≥50% Reduction from Baseline at Week 8 | Baseline and Week 8
  Blood samples will be collected at baseline and at Week 8 to assess the percentage of participants who have LDL-C <70 mg/dL and ≥50% reduction from baseline.
Percentage of Participants with LDL-C <55 mg/dL and ≥50% Reduction from Baseline at Week 8 | Baseline and Week 8
  Blood samples will be collected at baseline and at Week 8 to assess the percentage of participants who have LDL-C <55 mg/dL and ≥50% reduction from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (77):
- United States (35):
  - Central Research Associates ( Site 0009), Birmingham, Alabama
  - G&L Research ( Site 0024), Foley, Alabama
  - Synexus Clinical Research US, Inc. - Phoenix Central ( Site 0030), Phoenix, Arizona
  - Alliance for Multispecialty Research LLC ( Site 0049), Tempe, Arizona
  - Chemidox Clinical Trials ( Site 0008), Lancaster, California
  - Clinical Trials Research ( Site 0036), Sacramento, California
  - Legacy Clinical Trials ( Site 0044), Colorado Springs, Colorado
  - Alliance for Multispecialty Research, LLC ( Site 0040), Fort Myers, Florida
  - Soffer Health Institute ( Site 0046), Hollywood, Florida
  - East Coast Institute for Research ( Site 0041), Lake City, Florida
  - Inpatient Research Clinic ( Site 0017), Miami Lakes, Florida
  - Clinical Research Trials of Florida ( Site 0001), Tampa, Florida
  - Clinical Site Partners LLC, dba CSP Orlando ( Site 0014), Winter Park, Florida
  - Trialmed ( Site 0026), Chicago, Illinois
  - Great Lakes Clinical Trials - Ravenswood ( Site 0018), Chicago, Illinois
  - Midwest Institute For Clinical Research ( Site 0033), Indianapolis, Indiana
  - Alliance for Multispecialty Research, LLC ( Site 0048), Newton, Kansas
  - Cotton O'Neil Clinical Research Center ( Site 0006), Topeka, Kansas
  - L-MARC Research Center ( Site 0004), Louisville, Kentucky
  - Jubilee Clinical Research ( Site 0031), Las Vegas, Nevada
  - Cardiovascular Associates of the Delaware Valley ( Site 0035), Elmer, New Jersey
  - New Mexico Clinical Research & Osteoporosis Center, Inc. ( Site 0027), Albuquerque, New Mexico
  - Alliance for Multispecialty Research, LLC - Norman ( Site 0043), Norman, Oklahoma
  - Cardiology Consultants of Philadelphia Yardley ( Site 0016), Yardley, Pennsylvania
  - Provecta Research Network LLC ( Site 0022), Houston, Texas
  - Permian Research Foundation ( Site 0005), Odessa, Texas
  - LinQ Research ( Site 0025), Pearland, Texas
  - Clinical Trials of Texas, Inc. ( Site 0010), San Antonio, Texas
  - Stone Oak, LLC dba Discovery Clinical Trials (DCT) ( Site 0021), San Antonio, Texas
  - LinQ Research - Tomball ( Site 0047), Tomball, Texas
  - Conquest Research ( Site 0045), Arlington, Virginia
  - Manassas Clinical Research Center ( Site 0002), Manassas, Virginia
  - Health Research of Hampton Roads, Inc. ( Site 0013), Newport News, Virginia
  - National Clinical Research, Inc ( Site 0028), Richmond, Virginia
  - Rainier Clinical Research ( Site 0023), Renton, Washington
- Argentina (7):
  - CEMEDIC ( Site 0201), CABA, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 0202), Mar del Plata, Buenos Aires
  - CIPREC-CIPREC Sede Arenales ( Site 0200), Buenos Aires, Buenos Aires F.D.
  - Fundacion Estudios Clinicos ( Site 0203), Rosario, Santa Fe Province
  - Instituto de Investigaciones Clinicas Rosario ( Site 0204), Rosario, Santa Fe Province
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada ( Site 0206), CABA
  - Instituto de Cardiología "Juana F. Cabral"-Cardiología ( Site 0205), Corrientes
- Australia (6):
  - Australian Clinical Research Network ( Site 0900), Maroubra, New South Wales
  - Momentum Darlinghurst ( Site 0906), Sydney, New South Wales
  - Momentum Clinical Research Taringa ( Site 0907), Taringa, Queensland
  - Fusion Clinical Research ( Site 0901), Norwood, South Australia
  - Emeritus Research ( Site 0904), Camberwell, Victoria
  - Baker - HeartWest ( Site 0902), Hoppers Crossing, Victoria
- Brazil (5):
  - Centro de Pesquisas em Diabetes e Doenças Endócrino-Metabólicas ( Site 0306), Fortaleza, Ceará
  - Centro de Pesquisa Clinica do Coracao ( Site 0303), Aracaju, Sergipe
  - Hospital Universitário São Francisco de Assis - Bragança Paulista ( Site 0305), Bragança Paulista, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto ( Site 0309), São José do Rio Preto, São Paulo
  - IBPClin - Instituto Brasil de Pesquisa Clínica ( Site 0302), Rio de Janeiro
- Canada (5):
  - G A Research Associates ( Site 0102), Moncton, New Brunswick
  - Milestone Research Inc. ( Site 0111), London, Ontario
  - North York Diagnostic and Cardiac Centre ( Site 0110), North York, Ontario
  - Centricity Research Mirabel Multispecialty ( Site 0107), Mirabel, Quebec
  - Recherche Clinique Sigma Inc ( Site 0108), Québec, Quebec
- Hungary (4):
  - Lausmed Egészségügyi Szolgáltató ( Site 1105), Baja, Bács-Kiskun county
  - Borbánya Praxis ( Site 1103), Nyíregyháza, Szabolcs-Szatmár-Bereg
  - DRC Gyógyszervizsgáló Központ ( Site 1109), Balatonfüred, Veszprém megye
  - Debreceni Egyetem Klinikai Kozpont-Belgyógyászati Klinika (Anyagcsere Tanszék) ( Site 1102), Debrecen
- Israel (5):
  - Barzilai Medical Center ( Site 0504), Ashkelon
  - Linn Medical Center ( Site 0503), Haifa
  - Rambam Health Care Campus ( Site 0500), Haifa
  - Meir Medical Center. ( Site 0501), Kfar Saba
  - Clalit Health Services - Sakhnin Community Clinic ( Site 0502), Sakhnin
- Spain (2):
  - EAP Sardenya ( Site 0601), Barcelona
  - EBA Centelles ( Site 0600), Barcelona
- Turkey (Türkiye) (3):
  - Hacettepe Universite Hastaneleri ( Site 0700), Sıhhiye, Ankara
  - Eskisehir Osmangazi University ( Site 0705), Eskişehir
  - İnönü Üniversitesi Turgut Özal Tıp Merkezi ( Site 0702), Malatya
- United Kingdom (5):
  - Velocity Clinical Research Romford ( Site 0803), Bristol, Bristol, City of
  - West Walk Surgery ( Site 0801), Yate, Gloucestershire
  - Velocity Clinical Research Havering ( Site 0804), London, Havering
  - William Harvey Heart Centre ( Site 0800), London, London, City of
  - Lakeside Surgery ( Site 0802), Corby, Northamptonshire

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com